CLINICAL TRIAL: NCT01936857
Title: Buprenorphine to Improve HIV Care Engagement and Outcomes: A Randomized Trial (BRAVO)
Brief Title: Buprenorphine to Improve HIV Care Engagement and Outcomes
Acronym: BRAVO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Hanoi Medical University (Other); Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, P. Todd Korthuis, MD, Professor of Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA037441_VNE; 1R01DA037441 (NIH)
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Results first posted 2020-06-24 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: HIV; Substance Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Buprenorphine/naloxone (Experimental): Office based treatment of opioid dependence with buprenorphine/naloxone
  Interventions: Drug: Buprenorphine/naloxone
- Methadone Maintenance Therapy (Active Comparator): Referral to methadone maintenance therapy for treatment of opioid dependence.
  Interventions: Drug: Methadone Maintenance Therapy

INTERVENTIONS:
Drug: Buprenorphine/naloxone — Buprenorphine/naloxone induction begins with a 2-4mg test dose followed by additional doses on the day of induction to relieve withdrawal symptoms, and then titrated to a maintenance dose between 8-24 mg/day over 1 to 3 days. Doses will be directly observed and occur daily. After a minimum of 2 weeks, dosing may be changed to 3 or 4 times per week, as determined clinically appropriate by the HIV clinic study physician. Dosing will remain flexible to a maximum dose of 24mg for daily dosing and 32mg for every other day dosing, as deemed clinically appropriate by the study physician.
  Other Names: Suboxone
  Arms: Buprenorphine/naloxone
Drug: Methadone Maintenance Therapy — Subjects randomized to methadone maintenance therapy (MMT) referral will meet with an HIV clinic case manager who will facilitate referral to MMT. Methadone dosing will be managed by MMT staff, who dispense methadone according to Ministry of Health guidelines for MMT.
  Arms: Methadone Maintenance Therapy

SUMMARY:
The purpose of this study is to compare two models of substance abuse treatment in Vietnam, and how they each affect HIV care. In Vietnam, the current model for treating people with HIV who are also dependent on opioids is to refer them to methadone maintenance treatment centers. The new model the protocol will study is treatment of HIV and opioid dependence with buprenorphine/naloxone and counseling in the HIV clinic.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Current moderate or severe Diagnostic and Statistical Manual (DSM-V) opioid use disorder
* Urine drug screen positive for opioids
* Interested in receiving treatment for opioid dependence
* Age at least 18 years old
* Willing to practice an effective method of birth control, if female

Exclusion Criteria:

* Known hypersensitivity to buprenorphine or naloxone
* aspartate aminotransferase (AST) & alanine aminotransferase (ALT) > 5x upper limit
* Currently pregnant or breastfeeding
* Serious medical or psychiatric illness in past 30 days (e.g. opportunistic infection, psychosis) that precludes safe participation in the opinion of study physician
* Methadone maintenance treatment within 30 days of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip T Korthuis, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (6):
- Vietnam (6):
  - Bac Giang PAC OPC, Bắc Giang
  - Dong Da OPC, Hanoi
  - Hoang Mai HIV Clinic, Hanoi
  - Long Bien, Hanoi
  - Tu Liem, Hanoi
  - Thanh Hoa PAC OPC, Thanh Hóa

REFERENCES:
- [Derived] Edsall A, Hoffman KA, Thuy DT, Mai PP, Hang NT, Khuyen TT, Trang NT, Kunkel LE, Giang LM, Korthuis PT. Use of methamphetamine and alcohol among people with opioid use disorder and HIV in Vietnam: a qualitative study. BMC Public Health. 2021 Sep 22;21(1):1718. doi: 10.1186/s12889-021-11783-9. PMID 34548042
- [Derived] Korthuis PT, King C, Cook RR, Khuyen TT, Kunkel LE, Bart G, Nguyen T, Thuy DT, Bielavitz S, Nguyen DB, Tam NTM, Giang LM. HIV clinic-based buprenorphine plus naloxone versus referral for methadone maintenance therapy for treatment of opioid use disorder in HIV clinics in Vietnam (BRAVO): an open-label, randomised, non-inferiority trial. Lancet HIV. 2021 Feb;8(2):e67-e76. doi: 10.1016/S2352-3018(20)30302-7. PMID 33539760

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buprenorphine/Naloxone | Methadone Maintenance Therapy
Started | 141 | 140
Completed | 107 | 115
Not Completed | 34 | 25
Not completed — Sent to prison or 06 center | 11 | 12
Not completed — Lost to Follow-up | 10 | 7
Not completed — Death | 7 | 3
Not completed — Moved | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Side effect of medication | 1 | 0
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine/Naloxone | Methadone Maintenance Therapy | Total
Number analyzed (Participants) | 141 | 140 | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (5.8) | 38.6 (6.4) | 38.3 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 136 | 136 | 272
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Kinh | 139 | 139 | 278
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Vietnam | 141 | 140 | 281

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With HIV Viral Suppression
Description: HIV-1 RNA < 200 copies/mL
Time Frame: 12 months
Population: Follow up viral suppression was not available for 50 buprenorphine group participants, and 33 of methadone group participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine/Naloxone | Methadone Maintenance Therapy
Number analyzed (Participants) | 141 | 140
Participants
  Viral suppression at baseline: number analyzed (Participants) | 140 | 140
  Viral suppression at baseline | 97 | 92
  Viral suppression at 12 months: number analyzed (Participants) | 91 | 107
  Viral suppression at 12 months | 74 | 99

2. Primary Outcome: Participants With Heroin Use (Urine Drug Screen)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine/Naloxone | Methadone Maintenance Therapy
Number analyzed (Participants) | 98 | 110
Participants | 66 | 72

3. Primary Outcome: Participants With Heroin Use (Self-report)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine/Naloxone | Methadone Maintenance Therapy
Number analyzed (Participants) | 107 | 115
Participants | 64 | 67

4. Secondary Outcome: Number of Participants in Receipt of Antiretroviral Therapy (ART)
Description: Initiation of and retention on treatment with antiretroviral medications.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine/Naloxone | Methadone Maintenance Therapy
Number analyzed (Participants) | 128 | 131
Participants | 108 | 116

5. Secondary Outcome: Number of Participants in Retention in HIV Care
Description: HIV clinic visit in past 3 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine/Naloxone | Methadone Maintenance Therapy
Number analyzed (Participants) | 141 | 140
Participants | 111 | 118

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Buprenorphine/Naloxone | Methadone Maintenance Therapy
All-Cause Mortality (participants affected / at risk) | 7/141 | 3/140
Serious Adverse Events (participants affected / at risk) | 10/141 | 4/140
Other Adverse Events (participants affected / at risk) | 23/141 | 3/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine/Naloxone (N=141) | Methadone Maintenance Therapy (N=140)
Accident, trauma, or external factor (Injury, poisoning and procedural complications) | 6 (7) | 1 (1) — Includes overdose
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nephrogenic (Renal and urinary disorders) | 1 (1) | 0 (0)
AIDS-related (Immune system disorders) | 3 (3) | 2 (2)
(General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Psychiatric (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine/Naloxone (N=141) | Methadone Maintenance Therapy (N=140)
Unintentional injury (Injury, poisoning and procedural complications) | 12 (12) | 2 (2)
Abnormal lab result (General disorders) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Suspected infection (Infections and infestations) | 5 (5) | 0 (0)
Vascular (Vascular disorders) | 1 (1) | 0 (0)
Cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 4 (4) | 0 (0)
Headache (General disorders) | 2 (2) | 0 (0)
Allergic reaction (non-study medication) (Immune system disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT01936857/Prot_SAP_000.pdf